CLINICAL TRIAL: NCT06905184
Title: Activity PRN: Establishing Meaningful Occupation as and When Required Across Acute Inpatient Mental Health and Psychiatric Intensive Care Units
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cygnet Healthcare (Other)
Responsible Party: Principal Investigator, Neil Barker, Head of Occupational Therapy, Cygnet Healthcare
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Activity PRN
Record Dates: First submitted 2025-03-25; First posted 2025-04-01 (Actual); Last update posted 2025-04-01 (Actual); Status verified 2025-03

CONDITIONS: Activity Engagement
Keywords: Activity PRN; Occupational Therapy; Cygnet Healthcare; Mental Health; PICU; Acute
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: Treatment: One or more interventions are being evaluated for treating a disease, syndrome, or condition.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patient Group (Experimental): Individuals aged 18-65 years, admitted to a Psychiatric Intensive Care Unit or Acute Mental Health Unit, who receive the intervention Activity PRN.
  Interventions: Behavioral: Activity PRN

INTERVENTIONS:
Behavioral: Activity PRN — An Activity PRN plan will be delivered to consenting patients, as described above. The intervention will be communicated to them as a new approach that 'supports the individual to engage in personalised meaningful activities, which they can engage in as and when required'.
  Activity Resources are organised within a suitable, accessible location according with the patient's risk management and support plan. Dependent on the plan, resources may be kept on their person, in their bedroom, in a communal area, or in a locked or unlocked accessible cupboard.
  Ward staff will facilitate prn activities on an 'as and when required' basis. This can occur when: 1) a patient requests an activity from their card, 2) the patient appears disengaged, or 3) staff deem that the patient may benefit from participation in an activity for the purpose of engagement or distraction.

SUMMARY:
Design

A quasi-experimental mixed methods design research study will be conducted within:

Pippin Ward, a 10 bed Female PICU within Cygnet Appletree (data collected January - June 2022).

Haywood Ward, a 16 Male Acute within Cygnet Kewstoke. Nash Ward, a 12 bed Male PICU within Cygnet Kewstoke. Sandford Ward, a 16 bed Female Acute within Cygnet Kewstoke. Juniper Ward, a 17 bed Male Acute within Cygnet Churchill. Castle Ward, a 12 bed Female PICU within Cygnet Godden Green. Oakwood ward, a 15 bed Female Acute within Cygnet Godden Green.

The study will measure the change in provision of meaningful activity types, and frequency of participation within meaningful activities, as a result of the intervention, 'Activity PRN', on participating wards within Cygnet Healthcare Ltd.

Activity PRN, is an approach that uses occupational therapy approaches to facilitate meaningful activities as and when required. A 'prn activity' is any personally meaningful activity which can be facilitated as and when required, and is not a timetabled activity or session.

To show the effect of the intervention, a three month control period, pre-intervention, will measure the number of meaningful activity types provided, facilitated on an 'ad-hoc' basis, and participation frequency. A two week period will follow, in which ward based staff will receive training to implement Activity PRN. A further three month intervention period will measure the number of prn activity types provided, and the participation frequency of prn activities, as a result of delivering Activity PRN. It is hoped that about 60 patients will consent to receive the intervention.

DETAILED DESCRIPTION:
Ethical considerations All patients are invited to take part in the study, unless for any reason the Multi-Disciplinary Team decides that the patient is unsafe to take part, or cannot otherwise engage in meaningful activities on an as and when required basis.

Patients are selected to take part in the study by decision of their Multi-Disciplinary Team, that they have the capacity to make the decision to take part. At this point they are invited to read a Participant Information Sheet (appendix one), and given the opportunity to ask questions and clarify understanding of what the study involves and what they will need to do.

Patients are then asked to sign an Informed Consent Form (appendix two), to confirm understanding and that they agree to take part. A witness will also sign the form, who will be the occupational therapist or occupational therapy assistant on the ward. They have a right to withdraw their consent without affecting their rights as a patient.

After the informed consent form is signed, the patient is asked to contact their occupational therapist or occupational therapy assistant to start receiving the intervention, and a contact telephone and email for them is given on the patient information sheet.

Activity PRN is still offered as an intervention even if the patient declines to take part in the study.

Pre-Intervention To deliver the control intervention, Activity PRN is not implemented during an initial three month period. Patients however will have access to ad-hoc personally meaningful activities as part of a general ward environment. To maintain effect of the control period, neither ward staff nor patients will be made aware of the study.

To measure the number of ad-hoc meaningful activity types provided, and participation frequency, the following will be carried out:

* A therapeutic ward programme consisting of individual and group interventions will be delivered, as per standard practice.
* An occupational therapist, occupational therapy assistant or activity coordinator will take activity data from day and night shift documentation, in which activities are listed as per standard practice.
* A spreadsheet will be used to collect data (appendix three) of the description and number of meaningful activities engaged in by patients, and participation frequency of each meaningful activity.

Staff Training

A two-week break will take place following the pre-intervention to deliver staff training. As part of the training course, the following will take place:

The project manager facilitates training sessions using virtual technology, and where possible in house training until the whole ward team is trained. Nursing and support staff are supported to learn Activity PRN terminology, use the activity cards and engage service users in their prn activities, and record activity participation.

Intervention

To deliver Activity PRN as an intervention over a three month period, the following will be carried out:

* A therapeutic ward programme consisting of individual and group interventions will be delivered, as per standard practice.
* An Activity PRN plan will be delivered to consenting patients, as described above. The intervention will be communicated to them as a new approach that 'supports the individual to engage in personalised meaningful activities, which they can engage in as and when required'.
* Patients who do not consent are still eligible to receive access to any ad-hoc meaningful activity, as part of the normal ward environment, which will include any new activities added as part of implementing Activity PRN on the ward.
* An occupational therapist (or occupational therapy assistant or activity coordinator under the guidance of an occupational therapist) will gather information on patient interests using traditional methods.
* An occupational therapist (or occupational therapy assistant or activity coordinator under the guidance of an occupational therapist), will support patients to create an Activity PRN plan, by following the Activity PRN process (appendix four).
* Each activity must be a personally meaningful activity, accessible within a reasonable timeframe, and not a planned session within a therapeutic programme.
* Each activity is risk managed by a Multi-Disciplinary Team, and an appropriate support level is assigned, either independent, supervised or supported.
* Patient occupational function may also influence the support level assigned, or decision not to go ahead with the activity.
* Required activity resources are purchased according to need.
* Activity Resources are organised within a suitable, accessible location according with the patient's risk management and support plan. Dependent on the plan, resources may be kept on their person, in their bedroom, in a communal area, or in a locked or unlocked accessible cupboard.
* An Activity PRN plan is produced using a revised version of the Activity PRN card (appendix five). This will contain up to five personally meaningful prn activities. The card describes the support level required (independent, supervised or supported), resources, storage locations and activity locations in order to facilitate the activities. An activity log is included on the back of the card to record activity engagement.
* Ward staff will receive a copy of patient Activity PRN cards, as well as the patient receiving a personal card.
* Staff cards will be kept within the nursing station, within an 'Activity PRN Station', which is a document holder containing Activity PRN cards, and relevant signage drawing attention to staff and patients.
* Ward staff will facilitate prn activities on an 'as and when required' basis. This can occur when: 1) a patient requests an activity from their card, 2) the patient appears disengaged, or 3) staff deem that the patient may benefit from participation in an activity for the purpose of engagement or distraction.
* An occupational therapist may review the Activity PRN plan according to need.

To measure the number of prn activity types provided, and participation frequency, the following will be carried out:

* A therapeutic ward programme consisting of individual and group interventions will be delivered, as per standard practice.
* An occupational therapist (or occupational therapy assistant or activity coordinator under the guidance of an occupational therapist) will provide once daily support to nursing and ward staff, so that they continue to understand use of Activity PRN cards, and are able to continue to offer support to individuals.
* Activity PRN cards are checked daily to ensure recording is correct and kept up to date, and remain alongside observation records, so that continuous support can be offered to patients.
* Activity PRN cards are replaced if damaged beyond use, or the recording log is filled.
* An occupational therapist (or occupational therapy assistant or activity coordinator under the guidance of an occupational therapist) will collect activity data from the Activity PRN cards daily. This may include any additional prn activities recorded, which were not originally planned. Ward staff will be prompted to record the activities daily to maintain consistency of recording.
* A spreadsheet will be used to collect data (appendix three). This will be used to describe and calculate the number of prn activities, and participation frequency in each prn activity. Data on support level used, resources, storage and activity locations will also be collected, to provide additional information as a treatment resource guide for clinicians.

Data Processing

To process results, the following will be carried out:

* The total number of activities offered will be calculated across all participating sites, for the pre-intervention and intervention period.
* The total number of activities participated in will be calculated, for both study periods.
* A statistical analysis (ANOVA) will be run to compare the effect of the pre-intervention period and intervention period on the number of ad hoc meaningful activities and prn activities.
* A separate statistical analysis (ANOVA) will be run to compare the effect of the pre-intervention period and intervention period on participation frequency of ad hoc meaningful activities and prn activities.
* An additional independent variable is the number of participants between pre-intervention and post-intervention groups.

Study Limitations

* Activities that take place on an independent basis may not be observed by a member of staff in between observation periods, so this may reduce activity recording.
* Baseline data of ad hoc meaningful activities offered and participation frequency may differ between hospital sites, according to facilities and resources available, support levels given to patients and meaningful activity culture within the staff mix. This may impact on the data and affect statistical differences between the pre-intervention and post intervention periods.
* Some hospital sites may have different mixtures of occupational therapy staff, and may include one or both an occupational therapy assistant and activity coordinator. An occupational therapist will always be present.

ELIGIBILITY:
Inclusion Criteria:

Male or Female 18-65 Any ethnicity Any socio economic grouping Must be admitted to hospital for any primary diagnosis of a mental health condition Location as per units referred to in the study setting

Exclusion Criteria:

Excluded participants are those who do not give informed consent, or cannot give informed consent by review of the Multi-Disciplinary Team within participating wards.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-03-25 (Actual)

PRIMARY OUTCOMES:
PRN Activities | 6 months
  An increase in provision of 'as when required' (prn) activities across all services monitored.
Participation rate | 6 months
  An increase in participation frequency of 'prn activities', compared to 'ad hoc' meaningful activities pre-intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Cygnet Maidstone Hospital, Maidstone, Kent, United Kingdom

IPD SHARING:
Plan to Share IPD: No